CLINICAL TRIAL: NCT04187625
Title: Cell-based Therapy for the Treatment of Kidney Disease
Acronym: CTKD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003586
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Open label single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will be given autologous endothelial progenitor cells
  Interventions: Biological: endothelial progenitor cell

INTERVENTIONS:
Biological: endothelial progenitor cell — Kidney-derived endothelial progenitor cells will be delivered percutaneously to the kidney blood supply.

SUMMARY:
Endothelial progenitor cells derived from and delivered to the renal vasculature may be stimulated to initiate differentiation programs during episodes of injury. It is hypothesized that endothelial progenitor cells from the kidney can transition to a phenotype that promotes endothelial repair.

DETAILED DESCRIPTION:
This is an interventional study involving patients that have a diagnosis of chronic kidney disease. Patients will have at least stage 3 chronic kidney disease stage or greater. Kidney-derived endothelial progenitor cells will have been obtained using associated protocols that are currently approved by the Partners Human Research Committee.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients will have endothelial progenitor cells previously acquired.

Exclusion Criteria:

* Patients without previously acquired endothelial progenitor cells will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety of progenitor cell delivery | 180 days
  Serum creatinine will be measured after cell delivery

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Siedlecki, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Outcomes of individual participant data will be made available in a de-identified fashion.
Supporting Information: CSR
Time Frame: The clinical study report will be available at the conclusion of the study.
Access Criteria: Requests will be made to the study principal investigator.